CLINICAL TRIAL: NCT05639257
Title: Treatment of Myotonia - Lamotrigine Versus Namuscla
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grete Andersen, MD (Other)
Collaborators: GCP-Copenhagen (Unknown); Region Capital Denmark (Other); Danish Region (Unknown); Lupin Atlantis Holdings S.A. (Unknown); ZiteLab (Unknown)
Responsible Party: Sponsor-Investigator, Grete Andersen, MD, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-003784-94
Record Dates: First submitted 2022-10-04; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Non-Dystrophic Myotonia
Keywords: Becker myotonia; Thomsen myotonia; Paramyotonia; Hyperkalemic periodic paralysis
MeSH Terms: conditions — Paralysis, Hyperkalemic Periodic | interventions — Lamotrigine; Mexiletine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lamotrigine (Active Comparator): An escalation phase of 28 days:
  - tablet Lamotrigine 25 mg once daily in 14 days followed by 50 mg once daily in 14 days.
  A treatment phase of 30 days:
  - tablet Lamotrigine 100 mg, once daily in 10 days, twice daily in 10 days, followed by third daily in 10 days.
  Interventions: Drug: Lamotrigine
- Namuscla (Active Comparator): A placebo phase of 28 days:
  - tablet placebo 25 mg once daily in 14 days followed by 50 mg once daily in 14 days.
  A treatment phase of 30 days:
  - tablet Namuscla 167 mg, once daily in 10 days, twice daily in 10 days, followed by third daily in 10 days.
  Interventions: Drug: Namuscla

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine tablets increasing dosis to maximal 300 mg daily
  Arms: Lamotrigine
Drug: Namuscla — Namuscla tablets increasing dosis to maximal 501 mg daily
  Other Names: mexiletine
  Arms: Namuscla

SUMMARY:
In this clinical study, the aim is to investigate whether there is a difference in treatment of myotonia using two drugs. A difference there can justify the significantly higher cost when treated by Namuscla versus Lamotrigine.

According to the current corona pandemic, the investigators designed an app to use for data collection in the study. The app also ensures that patients who live far from the clinic more easily can participate.

DETAILED DESCRIPTION:
On 18 May 2020, the National Board of Health in Denmark approved Namuscla for the treatment of myotonia. Myotonia is a congenital muscle disease that delays muscle relaxation after a muscle contraction. Myotonia can be disabling, but with treatment, most are able to work. Namuscla is the first registered drug to treat myotonia, however, the active part mexiletine is not new. It has been used off-label to treat myotonia for decades. The price for the new preparation is high with a daily cost (approx. 70 EU/dollar). In 2017, the investigators found evidence that treatment with lamotrigine is efficacious against myotonia. Treatment with lamotrigine can reduce the price to 150 EU/dollar per year.

Therefore, the aim of the study is to investigate whether there is a difference in the effects om myotonia and side effects of the two drugs, which can justify the significantly higher cost when treated with Namuscla in a double blinded, inferiority, cross-over study lasting 4 months.

According to the current corona pandemic, the study is designed without need of physical attendance so that inclusion and collection of experimental data can take place, by phone conversations, video-guided testing, and diary registration via a study-App. It also ensures that patients who live far away more easily can participate. Blood tests and ECGs can be performed locally.

ELIGIBILITY:
Inclusion Criteria:

1. Capable adult women and men (age ≥ 18 years).
2. Diagnosed with Myotonia Congenita (Becker and Thomsen type), Paramyotonia Congenita, or Hyperkalemic periodic paralysis.
3. Myotonia under treatment or which significantly limits the daily activities (MBS> 2).

Exclusion Criteria:

1. Allergy to lamotrigine, mexiletine, or the inactive ingredients in trial medication.
2. Disease, which is affected by trial medication such as heart disease (ischemia and arrhythmia), epilepsy, and significant renal or hepatic failure.
3. Treatment that, in the opinion of the project manager, can affect the study result - medication with significant interactions with trial medication.
4. In case of smoking, start or cessation during the study.
5. Pregnant or breastfeeding during the study period. Fertile women with a positive pregnancy test at the time of entry into the trial, or who do not use safe contraception during the project period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Myotonia Behavior Scale (MBS) | baseline and week 8
  Each participant chose one of six statements about how myotonia affect their daily living. MBS is register once daily in a week. 1 is no symptoms of myotonia, 6 is invalidating symptoms of myotonia.
  Measured without treatment and in the last week of treatment.

SECONDARY OUTCOMES:
Change in Eye-myotonia | baseline and week 8
  Eye opening test (time in seconds): Eyes are pinched with maximum strength for 5 sec, then opened ASAP. Repeated 5 times. Longer times measured more server myotonia in eye muscles.
Change in hand-myotonia | baseline and week 8
  Hand opening test (time in seconds): Right hand is closed with maximum strength for five seconds before opened as soon as possible. Time is measured in seconds. Longer times measured more server myotonia in hand muscles. Repeated 5 times.
Change in time-up-and-go-test (TUG) | baseline and week 8
  TUG - time-up&go (time in seconds): After 10 minutes rest in a chair, participants get up, walk 3 meters, turn around, returning to the chair performed in regular pace. Longer times measured more server myotonia in legs muscles.
Change in Individualized Neuromuscular Quality of Life Questionnaire (INQoL) | baseline and week 8
  A questionnaire for patients with neuromuscular diseases measuring quality of life and the impact of the disease on everyday life. The INQoL is composed of 45 items investigating 4 dimensions, subdivided into 11 sub-dimensions. The scoring of the INQoL generates a profile (0-100). Higher score scores = higher impact of disorders. The form is translated in Danish.
Days with Side effects (SE) | through study completion, in total 123 days
  Side effects are noted daily. Participants have three opportunities they can 1) cross no SE, 2) cross a specific SE on an alphabetically list containing all known SE for both drugs, or 3) they can describe a AE under other.
Change in Side Effect Scale (SE) | baseline and week 8
  Each participant chose one of six statements about how side effects affect their daily living. SES is register once daily in a week. 1 is no side effects, 6 is invalidating side effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, department of Neurology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No